CLINICAL TRIAL: NCT06971367
Title: Transformative Approaches to Rapidly and Efficiently Test Demand Creation Interventions to Promote HIV Retesting in Adults at Increased Risk of HIV
Brief Title: IBIS Megastudy of Interventions to Encourage HIV Retesting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Pennsylvania (Other); Kenya Medical Research Institute (Other); Infectious Diseases Research Collaboration, Uganda (Other); University of California, Berkeley (Other); Makerere University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 23-39197- 2; R01MH132438 (NIH)
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: HIV
Keywords: behavioral economics; "nudge" interventions; megastudy; Uganda; Kenya; HIV retesting

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- HIV risk assessment (Experimental): A message that adheres to the following core concepts: - Emphasize that a negative test doesn't mean that previous behavior(s) weren't high-risk - Enable people to re-assess their own personal risk at a later/future date - Suggest risk behaviors to reflect on - If participant has engaged in one or more behaviors, emphasize their need to re-test
  Interventions: Behavioral: Risk assessment messaging
- U=U messaging (Experimental): A message that adheres to the following core concepts: Explain benefits of finding out your HIV-positive status as early after infection as possible and start treatment as soon as possible. These benefits include: -Prevent transmission of HIV to anyone -Live a normal life, with freedom in sexual choices and ability to start a family
  Interventions: Behavioral: U=U messaging
- Community benefits (Experimental): A message that adheres to the following core concepts: - Emphasize that regular testing keeps the participant's community safe and healthy by reducing chances of transmitting HIV unknowingly - Call for responsibility- the participant to do their part for the community; they are an integral part of the solution
  Interventions: Behavioral: Community benefits messaging
- Fresh start effect (Experimental): A message that adheres to the following core concepts: - Using a specific moment in time (in this case, a negative HIV test) to motivate a healthy behavior (i.e. a "fresh start" moment) - emotional unburdening of resolving uncertainty (not knowing one's status is more stressful than knowing one's status, whether positive or negative, and being able to take healthy steps after knowing if the status is negative or positive)
  Interventions: Behavioral: Fresh start effect
- Education-based (Experimental): A message that adheres to the following core concepts: -Increase attention to HIV re-testing reminder through interactive trivia questions -Correct or reinforce understanding about HIV prevention, transmission, and retesting
  Interventions: Behavioral: Education-based messaging
- Default appointment (Experimental): A message that adheres to the following core concepts: - Having a set appointment will reduce uncertainty about availability for retest visit - Having an opt-out option for the future retesting appointment - A planning prompt to be specific about the participant's future plan for retesting - Gentle/soft commitment: by picking a date, mentally agree to come back to retest
  Interventions: Behavioral: Default appointment messaging
- "Reserved for you" (Experimental): A message that adheres to the following core concepts: - Make participant aware that the test is available, and the clinic is welcoming the participant to receive it - "VIP status-" the participant is lucky/special to have this opportunity
  Interventions: Behavioral: Reserved for you messaging
- Social norms- default messenger (Experimental): A message that adheres to the following core concepts: - Reduce stigma and normalize retesting by explaining that it is a common practice for people to be aware of their HIV status and get tested - Leverages social pressure to participate in retesting - Uses a relatable community member to deliver the message. Message delivered by the default avatar.
  Interventions: Behavioral: Social norms (default) messaging
- Social norms- varied messenger (Experimental): A message that adheres to the following core concepts: - Reduce stigma and normalize retesting by explaining that it is a common practice for people to be aware of their HIV status and get tested often when they are at risk - Leverages social pressure to participate in retesting - Uses a relatable community member to deliver the message. Message delivered by avatar that approximately matches the participant's age and sex
  Interventions: Behavioral: Social norms (varied) messaging
- Goal-setting (Experimental): A message that adheres to the following core concepts: -Encouraging motivation of participants to set a goal for follow-up testing -Empowering individuals through promotion of HIV retesting
  Interventions: Behavioral: Goal-setting messaging
- Incentive (Experimental): Participants receive a small financial incentive for returning for a repeat HIV test within 3-6 months from enrollment
  Interventions: Behavioral: Incentive
- Standard of care (Control) (No Intervention): Participants will receive standard of care messaging provided by Ministry of Health (MoH) HIV testing counselors.

INTERVENTIONS:
Behavioral: Risk assessment messaging — Participants will be shown a brief video message at their baseline visit, containing information related to HIV risk assessment core concepts and encouraging them to return for a repeat HIV test. They will also receive brief SMS follow-up messages at about 8 and 11 weeks after baseline reminding them about HIV retesting and re-emphasizing concepts from the HIV risk assessment content category.
  Arms: HIV risk assessment
Behavioral: U=U messaging — Participants will be shown a brief video message at their baseline visit, containing information related to U=U core concepts and encouraging them to return for a repeat HIV test. They will also receive brief SMS follow-up messages at about 8 and 11 weeks after baseline reminding them about HIV retesting and re-emphasizing concepts from the U=U content category.
  Arms: U=U messaging
Behavioral: Community benefits messaging — Participants will be shown a brief video message at their baseline visit, containing information related to Community Benefits core concepts and encouraging them to return for a repeat HIV test. They will also receive brief SMS follow-up messages at about 8 and 11 weeks after baseline reminding them about HIV retesting and re-emphasizing concepts from the Community Benefits content category.
  Arms: Community benefits
Behavioral: Fresh start effect — Participants will be shown a brief video message at their baseline visit, containing information related to Fresh Start core concepts and encouraging them to return for a repeat HIV test. They will also receive brief SMS follow-up messages at about 8 and 11 weeks after baseline reminding them about HIV retesting and re-emphasizing concepts from the Fresh start effect content category.
  Arms: Fresh start effect
Behavioral: Education-based messaging — Participants will be shown a brief video message at their baseline visit, containing information related to HIV education core concepts and encouraging them to return for a repeat HIV test. They will also receive brief SMS follow-up messages at about 8 and 11 weeks after baseline reminding them about HIV retesting and re-emphasizing concepts from the Education-based content category.
  Arms: Education-based
Behavioral: Default appointment messaging — Participants will be shown a brief video message at their baseline visit, containing information related to Default Appointment core concepts and encouraging them to return for a repeat HIV test. They will also receive brief SMS follow-up messages at about 8 and 11 weeks after baseline reminding them about HIV retesting and re-emphasizing concepts from the Default Appointment content category.
  Arms: Default appointment
Behavioral: Reserved for you messaging — Participants will be shown a brief video message at their baseline visit, containing information related to the "Reserved for you" core concepts and encouraging them to return for a repeat HIV test. They will also receive brief SMS follow-up messages at about 8 and 11 weeks after baseline reminding them about HIV retesting and re-emphasizing concepts from the "Reserved for you" content category.
  Arms: "Reserved for you"
Behavioral: Social norms (default) messaging — Participants will be shown a brief video message at their baseline visit, containing information related to Social Norms core concepts and encouraging them to return for a repeat HIV test. The video message will be delivered by the default avatar. They will also receive brief SMS follow-up messages at about 8 and 11 weeks after baseline reminding them about HIV retesting and re-emphasizing concepts from the Social Norms content category.
  Arms: Social norms- default messenger
Behavioral: Social norms (varied) messaging — Participants will be shown a brief video message at their baseline visit, containing information related to Social Norms core concepts and encouraging them to return for a repeat HIV test. The video message will be delivered by an avatar that approximately matches each participant's age and sex. They will also receive brief SMS follow-up messages at about 8 and 11 weeks after baseline reminding them about HIV retesting and re-emphasizing concepts from the Social Norms content category.
  Arms: Social norms- varied messenger
Behavioral: Goal-setting messaging — Participants will be shown a brief video message at their baseline visit, containing information related to goal-setting core concepts and encouraging them to return for a repeat HIV test. They will also receive brief SMS follow-up messages at about 8 and 11 weeks after baseline reminding them about HIV retesting and re-emphasizing concepts from the goal-setting content category.
  Arms: Goal-setting
Behavioral: Incentive — Participants will be informed that they will receive a small financial incentive if they return for repeat HIV testing in 3-6 months after enrollment.
  Arms: Incentive

SUMMARY:
In this study, the investigators will test the effectiveness of multiple low-cost behavioral interventions, designed with end-user input, to promote HIV retesting among adults in rural Kenya and Uganda who have higher risk of HIV exposure.

DETAILED DESCRIPTION:
HIV re-testing is crucial in ensuring early identification of disease to promote well-being of an individual as well as preventing onward spread of infection. The IBIS megastudy of interventions to encourage HIV retesting aims to test up to 12 different strategies aimed at encouraging repeat testing of HIV among individuals >/= 15 years old who are at increased risk of HIV infection. The different strategies are aimed at modifying individual behavior to enhance HIV testing. The study aims to enroll 30,000-40,000 individuals from 8 HIV testing sites in South West Uganda and Western Kenya. The study will then evaluate the effectiveness of the interventions by comparing HIV retesting rates 3-6 months later in the different study arms. The data collected during the study will further be used to understand which of the interventions offered worked best and for whom.

ELIGIBILITY:
Inclusion Criteria:

* at least 15 years of age
* Accessing HIV testing services at study-associated hospitals or clinics
* At increased risk of HIV infection (defined by national (Kenya or Uganda) MoH criteria)
* Documented negative HIV antibody test at time of enrollment
* No intent to migrate out of community in next 3 months
* Daily access to a mobile phone (required since some of the interventions will be delivered by phone)

Exclusion Criteria:

* HIV-positive at time of enrollment

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40000 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
HIV retesting uptake | Measured 3-6 months after baseline visit
  The proportion of participants in each study arm who return for repeat HIV testing within 3-6 months after the baseline visit.

SECONDARY OUTCOMES:
PrEP uptake at follow up | 3-6 months
  The proportion of participants who initiate PrEP at the time of HIV retesting, among those who are HIV-negative and not currently taking PrEP. PrEP dispensing will be done in accordance with Kenyan and Ugandan guidelines. Uptake will be recorded on study CRFs.

OTHER OUTCOMES:
HIV seroconversion at follow-up | Measured 3-6 months after baseline
  The proportion of participants returning for follow up who have a newly positive HIV test result. HIV seroconversion will be measured as documented rapid HIV antibody test at the time of study follow-up retesting (3-6 months after baseline).
Linkage to ART among those who seroconvert at follow-up | 3-6 months
  The proportion of participants that seroconvert at follow up who link to ART. ART dispensing will be done in accordance with Kenyan and Ugandan guidelines. Uptake will be recorded on study CRFs.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Chamie, MD, MPH, Principal Investigator — University of California, San Francisco; Harsha Thirumurthy, PhD, Principal Investigator — University of Pennsylvania
Locations (2):
- Kenya Medical Research Institution (KEMRI), Mbita, Kenya
- Infectious Diseases Research Collaboration (IDRC), Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share de-identified IPD from our baseline and follow-up questionnaires, which includes questions about subject demographics and HIV risk.
Supporting Information: Study Protocol
Time Frame: Data requests can be submitted starting 3 months after article publication and the data will be made accessible for up to 36 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP).